CLINICAL TRIAL: NCT02017717
Title: A Randomized Phase 3 Open Label Study of Nivolumab Versus Bevacizumab and Multiple Phase 1 Safety Cohorts of Nivolumab or Nivolumab in Combination With Ipilimumab Across Different Lines of Glioblastoma
Brief Title: A Study of the Effectiveness and Safety of Nivolumab Compared to Bevacizumab and of Nivolumab With or Without Ipilimumab in Glioblastoma Patients
Acronym: CheckMate 143
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-143; 2013-003738-34 (EudraCT Number)
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Results first posted 2022-06-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Nivolumab; Bevacizumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm N:Nivolumab (Experimental): Cohort 1, 1c, 1d and 2: Nivolumab specified dose on specified days
  Interventions: Biological: Nivolumab
- Arm N + I:Nivolumab + Ipilimumab (Experimental): Cohort 1: Nivolumab specified dose on specified days + Ipilimumab specified dose on specified days, then Nivolumab specified dose on specified days
  Cohort 1b: Nivolumab specified dose on specified days + Ipilimumab specified dose on specified days, then Nivolumab specified dose on specified days
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm B: Bevacizumab (Active Comparator): Cohort 2: Bevacizumab specified dose on specified days
  Interventions: Biological: Bevacizumab

INTERVENTIONS:
Biological: Nivolumab — specified dose on specified days
  Other Names: BMS-936558
  Arms: Arm N + I:Nivolumab + Ipilimumab; Arm N:Nivolumab
Biological: Bevacizumab — specified dose on specified days
  Other Names: Avastin
  Arms: Arm B: Bevacizumab
Biological: Ipilimumab — specified dose on specified days
  Other Names: Yervoy
  Arms: Arm N + I:Nivolumab + Ipilimumab

SUMMARY:
The purpose of the study is to compare the efficacy and safety of nivolumab administered alone versus bevacizumab in patients diagnosed with recurrent glioblastoma (a type of brain cancer, also known as GBM), and to evaluate the safety and tolerability of nivolumab administered alone or in combination with ipilimumab in patients with different lines of GBM therapy.

DETAILED DESCRIPTION:
Allocation: Randomized (Cohorts 1, 2 and Part B of 1c/1d), Non-Randomized (Cohorts 1b, and Part A of 1c/1d)

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed Grade IV malignant glioma
* Previous treatment with radiotherapy and temozolomide (Cohorts 1, 1b and 2 only)
* First recurrence of GBM (Cohorts 1, 1b and 2 only)
* First diagnosis of GBM with resectable disease (Cohorts 1c Part A only)
* First diagnosis of unmethylated MGMT GBM (Cohort 1d and Cohort 1c Part B only)
* Karnofsky performance score of 70 or higher

Exclusion Criteria:

* More than 1 recurrence of GBM (Cohorts 1, 1b and 2 only)
* Any recurrence of GBM (Cohorts 1c and 1d only)
* Presence of extracranial metastatic or leptomeningeal disease
* Active, known or suspected autoimmune disease
* Clinically significant cardiovascular disease
* Prior bevacizumab or other Vascular Endothelial Growth Factor (VEGF) or anti-angiogenic treatment (Cohort 2 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2014-02-07 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (108):
- United States (45):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - Local Institution - 0055, Los Angeles, California
  - Local Institution - 0009, Los Angeles, California
  - UCLA Neuro-Oncology Program, Los Angeles, California
  - Local Institution - 0014, San Francisco, California
  - The Regents of the University of California, San Francisco, San Francisco, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - Local Institution - 0021, Aurora, Colorado
  - Local Institution - 0001, New Haven, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Local Institution - 0002, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Local Institution - 0008, Baltimore, Maryland
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Local Institution - 0006, Boston, Massachusetts
  - Local Institution - 0043, Boston, Massachusetts
  - Local Institution - 0056, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Local Institution - 0003, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Local Institution - 0007, Durham, North Carolina
  - Preston Robert Tisch Brain Tumor Center at Duke University, Durham, North Carolina
  - Local Institution - 0049, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University - Clinical Research Institute, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Local Institution - 0023, Charleston, South Carolina
  - Medical University Of South Carolina, Charleston, South Carolina
  - Local Institution - 0005, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Local Institution - 0024, Houston, Texas
  - University Of Texas Md Anderson Cancer Ctr, Houston, Texas
  - University Of Virginia Health System, Charlottesville, Virginia
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
  - Local Institution - 0020, Seattle, Washington
  - Swedish Neuroscience Institute, Seattle, Washington
- Australia (8):
  - Local Institution - 0035, Liverpool, New South Wales
  - Local Institution, Liverpool, New South Wales
  - Local Institution - 0034, East Bentleigh, Victoria
  - Local Institution, East Bentleigh, Victoria
  - Local Institution - 0033, Heidelberg, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution - 0032, Nedlands, Western Australia
  - Local Institution, Nedlands, Western Australia
- Belgium (3):
  - Local Institution - 0050, Brussels
  - Local Institution, Brussels
  - Local Institution - 0051, Brussels
- Denmark (4):
  - Aarhus University Hospital, Aarhus C
  - Local Institution - 0058, Aarhus C
  - Local Institution - 0057, Odense C
  - Odense University Hospital, Odense C
- France (7):
  - Local Institution - 0062, Bron
  - Local Institution, Bron
  - Local Institution - 0063, Marseille
  - Local Institution, Marseille
  - Local Institution - 0068, Paris
  - Local Institution, Paris
  - Local Institution - 0064, Paris
- Germany (8):
  - Local Institution - 0037, Bonn
  - Universitaetsklinikum Bonn, Bonn
  - Klinikum Der J. W. Goethe-Universitaet Frankfurt/Main, Frankfurt am Main
  - Local Institution - 0036, Frankfurt am Main
  - Local Institution - 0038, Heidelberg
  - Local Institution, Heidelberg
  - Local Institution - 0041, Münster
  - Universitaetsklinikum Muenster, Münster
- Italy (8):
  - Local Institution - 0010, Bologna
  - Local Institution, Bologna
  - Local Institution - 0011, Milan
  - Local Institution, Milan
  - Local Institution - 0012, Siena
  - Local Institution, Siena
  - Azienda Ospedaliera Citta della Salute e della Scienza, Torino
  - Local Institution - 0013, Torino
- Netherlands (4):
  - Local Institution - 0067, Amsterdam
  - Local Institution, Amsterdam
  - Local Institution - 0066, Groningen
  - Local Institution, Groningen
- Poland (4):
  - Local Institution - 0060, Gdansk
  - Local Institution, Gdansk
  - Local Institution - 0059, Warsaw
  - Local Institution, Warsaw
- Spain (7):
  - Local Institution - 0047, Barcelona
  - Local Institution, Barcelona
  - Local Institution - 0045, Madrid
  - Local Institution, Madrid
  - Local Institution - 0046, Madrid
  - Local Institution - 0070, Pamplona
  - Local Institution, Pamplona
- Switzerland (4):
  - Centre hospitalier universitaire Vaudois (CHUV), Lausanne
  - Local Institution - 0039, Lausanne
  - Local Institution - 0040, Zurich
  - UniversitaetsSpital Zurich, Zurich
- United Kingdom (6):
  - Local Institution - 0018, London, Greater London
  - Local Institution, London, Greater London
  - Local Institution - 0015, Manchester, Greater Manchester
  - Local Institution, Manchester, Greater Manchester
  - Local Institution - 0017, Liverpool
  - Local Institution, Liverpool

REFERENCES:
- [Derived] de Melo SM, Elias Nunes da Silva ME, Torloni MR, Riera R, De Cicco K, Latorraca CO, Pinto ACPN. Anti-PD-1 and anti-PD-L1 antibodies for glioma. Cochrane Database Syst Rev. 2025 Jan 8;1(1):CD012532. doi: 10.1002/14651858.CD012532.pub2. PMID 39777725
- [Derived] Woroniecka K, Fecci PE. Immuno-synergy? Neoantigen vaccines and checkpoint blockade in glioblastoma. Neuro Oncol. 2020 Sep 29;22(9):1233-1234. doi: 10.1093/neuonc/noaa170. No abstract available. PMID 32691060
- [Derived] Reardon DA, Brandes AA, Omuro A, Mulholland P, Lim M, Wick A, Baehring J, Ahluwalia MS, Roth P, Bahr O, Phuphanich S, Sepulveda JM, De Souza P, Sahebjam S, Carleton M, Tatsuoka K, Taitt C, Zwirtes R, Sampson J, Weller M. Effect of Nivolumab vs Bevacizumab in Patients With Recurrent Glioblastoma: The CheckMate 143 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Jul 1;6(7):1003-1010. doi: 10.1001/jamaoncol.2020.1024. PMID 32437507
- [Derived] Stupp R. Drug development for glioma: are we repeating the same mistakes? Lancet Oncol. 2019 Jan;20(1):10-12. doi: 10.1016/S1470-2045(18)30827-1. Epub 2018 Dec 3. No abstract available. PMID 30522968
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 529 participants participated in the study. Of these 529 participants, 448 were randomized in the pre-treatment phase while 81 were directly treated in a non-randomized fashion. Of the 448 participants randomized, 423 moved to the treatment phase. The total number of treated participants was 504 (81 directly treated, 423 randomized and treated).
  GBM = Glioblastoma MGMT = O6-methylguanin-DNA-methyltransferase
Groups:
- Cohort 1: Arm N1+I3: Nivolumab 1 mg/kg administered as a 60-minute intravenous (IV) infusion followed by ipilimumab 3 mg/kg 90-minute IV infusion every 3 weeks for 4 cycles, then nivolumab 3 mg/kg 60-minute IV every 2 weeks thereafter
- Cohort 1: Arm N3; Cohort 2: Arm N3: Nivolumab 3 mg/kg dosed as 60-minute IV infusion every 2 weeks
- Cohort 1b: Arm N3+I1: Nivolumab 3 mg/kg administered as a 60-minute IV infusion followed by ipilimumab 1 mg/kg 90-minute IV infusion every 3 weeks for 4 cycles, then nivolumab 3 mg/kg 60-minute IV every 2 weeks thereafter
- Part A Cohort 1c: Arm N3+RT+TMZ; Part B Cohort 1c: Arm N3+RT+TMZ: Participants with newly diagnosed GBM: Nivolumab 3 mg/kg dosed as 60-minute IV infusion every 2 weeks with standard of care treatment including surgical resection and chemoradiation followed by 6 or more cycles of maintenance temozolomide
- Part A Cohort 1d: Arm N3+RT; Part B Cohort 1d: Arm N3+RT: Participants with newly diagnosed unmethylated MGMT GBM: Nivolumab 3 mg/kg dosed as 60-minute IV infusion every 2 weeks with standard of care treatment including surgical resection and radiation therapy
- Cohort 2: Arm B: Bevacizumab 10 mg/kg dosed every 2 weeks as 90-minute IV infusion for the first dose and 60-minute IV infusions for subsequent doses if the first infusion is tolerated
Period: Before Treatment Period
Arm/Group | Cohort 1: Arm N1+I3 | Cohort 1: Arm N3 | Cohort 1b: Arm N3+I1 | Part A Cohort 1c: Arm N3+RT+TMZ | Part A Cohort 1d: Arm N3+RT | Part B Cohort 1c: Arm N3+RT+TMZ | Part B Cohort 1d: Arm N3+RT | Cohort 2: Arm N3 | Cohort 2: Arm B
Started | 10 | 10 | 20 | 31 | 30 | 29 | 30 | 184 | 185
Randomized | 10 | 10 | 0 | 0 | 0 | 29 | 30 | 184 | 185
Completed (Completed = Moved to treatment period) | 10 | 10 | 20 | 31 | 30 | 28 | 28 | 182 | 165
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 20
Not completed — Adverse Event unrelated to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant request to stop therapy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Participant withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 11
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant no longer met criteria | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Not completed — other reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period
Arm/Group | Cohort 1: Arm N1+I3 | Cohort 1: Arm N3 | Cohort 1b: Arm N3+I1 | Part A Cohort 1c: Arm N3+RT+TMZ | Part A Cohort 1d: Arm N3+RT | Part B Cohort 1c: Arm N3+RT+TMZ | Part B Cohort 1d: Arm N3+RT | Cohort 2: Arm N3 | Cohort 2: Arm B
Started (Started = Treated) | 10 | 10 | 20 | 31 | 30 | 28 | 28 | 182 | 165
Completed (Completed = Continuing in the treatment period) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 10 | 20 | 31 | 30 | 28 | 28 | 182 | 165
Not completed — Disease progression | 7 | 9 | 12 | 20 | 26 | 16 | 22 | 165 | 135
Not completed — Study drug toxicity | 3 | 0 | 1 | 4 | 4 | 5 | 3 | 7 | 11
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse event unrelated to study drug | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 4 | 5
Not completed — Participant request to stop therapy | 0 | 0 | 3 | 6 | 0 | 2 | 1 | 4 | 7
Not completed — Participant withdrew consent | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 4
Not completed — Participant no longer met criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other reasons | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Not completed — Maximum clinical benefit | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Not reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cohorts 1b and 1c/1d (Part A) baseline characteristics are in regards to Treated Participants, while Cohorts 1, 1c/1d (Part B) and 2 baseline characteristics are in regards to Randomized Participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Arm N1+I3 | Cohort 1: Arm N3 | Cohort 1b: Arm N3+I1 | Part A Cohort 1c: Arm N3+RT+TMZ | Part A Cohort 1d: Arm N3+RT | Part B Cohort 1c: Arm N3+RT+TMZ | Part B Cohort 1d: Arm N3+RT | Cohort 2: Arm N3 | Cohort 2: Arm B | Total
Number analyzed (Participants) | 10 | 10 | 20 | 31 | 30 | 29 | 30 | 184 | 185 | 529
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (11.3) | 58.6 (10.9) | 55.0 (11.9) | 56.5 (11.3) | 58.2 (10.2) | 57.3 (12.7) | 58.8 (10.5) | 55.0 (11.3) | 54.2 (10.7) | 55.4 (11.1)
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 7 | 6 | 17 | 23 | 22 | 22 | 19 | 142 | 156 | 414
  >= 65 | 3 | 4 | 3 | 8 | 8 | 7 | 11 | 42 | 29 | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 6 | 11 | 8 | 10 | 9 | 68 | 66 | 187
  Male | 6 | 5 | 14 | 20 | 22 | 19 | 21 | 116 | 119 | 342
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 4 | 1 | 10
  Not Hispanic or Latino | 10 | 10 | 20 | 29 | 27 | 28 | 29 | 86 | 88 | 327
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 94 | 96 | 192
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race only
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Asian | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 7
    Black or African American | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 8
    White | 10 | 8 | 18 | 26 | 28 | 27 | 28 | 176 | 181 | 502
    Other | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 4 | 1 | 10
    Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-Related Adverse Events Leading to Discontinuation by Worst CTC Grade for All Treated Participants in Cohorts 1, 1b, 1c and 1d Who Permanently Discontinued Study Medication Prior to Completing Four Doses
Description: The percentage of participants who experienced a drug-related adverse event leading to drug discontinuation by worst grade (grade 5 being the worst) prior to complete four-dose treatment. Toxicities were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. MedDRA Version: 24.1
Time Frame: Includes events reported between first dose and 30 days after last dose of study therapy (up to 3 doses, up to approximately 2 months)
Population: All Treated Participants in Cohorts 1, 1b, 1c and 1d Who Permanently Discontinued Study Medication Prior to Completing Four Doses
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Arm N1+I3 | Cohort 1: Arm N3 | Cohort 1b: Arm N3+I1 | Part A Cohort 1c: Arm N3+RT+TMZ | Part A Cohort 1d: Arm N3+RT | Part B Cohort 1c: Arm N3+RT+TMZ | Part B Cohort 1d: Arm N3+RT
Number analyzed (Participants) | 6 | 4 | 7 | 3 | 1 | 4 | 4
Percentage of participants
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 16.7 | 0 | 0 | 66.7 | 0 | 0 | 50.0
  Grade 4 | 33.3 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Adverse Events (Worst Grade) in Cohorts 1, 1b, 1c and 1d
Description: The percentage of participants who experienced an adverse event by worst grade in each treatment arm. Toxicities were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. MedDRA Version: 24.1
Time Frame: From first dose to 30 days post last dose (up to approximately 34 months).
Population: All Treated Participants in Cohorts 1, 1b, 1c and 1d
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Arm N1+I3 | Cohort 1: Arm N3 | Cohort 1b: Arm N3+I1 | Part A Cohort 1c: Arm N3+RT+TMZ | Part A Cohort 1d: Arm N3+RT | Part B Cohort 1c: Arm N3+RT+TMZ | Part B Cohort 1d: Arm N3+RT
Number analyzed (Participants) | 10 | 10 | 20 | 31 | 30 | 28 | 28
Percentage of participants
  Grade 1 | 0 | 20.0 | 5.0 | 6.5 | 13.3 | 3.6 | 17.9
  Grade 2 | 10.0 | 30.0 | 25.0 | 12.9 | 26.7 | 28.6 | 25.0
  Grade 3 | 70.0 | 40.0 | 50.0 | 58.1 | 33.3 | 50.0 | 35.7
  Grade 4 | 20.0 | 10.0 | 20.0 | 22.6 | 20.0 | 10.7 | 21.4
  Grade 5 | 0 | 0 | 0 | 0 | 3.3 | 3.6 | 0

3. Primary Outcome: Percentage of Participants With Serious Adverse Events (Worst Grade) in Cohorts 1, 1b, 1c and 1d
Description: The percentage of participants who experienced a serious adverse event by worst grade in each treatment arm. Toxicities were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. MedDRA Version: 24.1
Time Frame: From first dose to 30 days post last dose (up to approximately 34 months).
Population: All Treated Participants in Cohorts 1, 1b, 1c and 1d
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Arm N1+I3 | Cohort 1: Arm N3 | Cohort 1b: Arm N3+I1 | Part A Cohort 1c: Arm N3+RT+TMZ | Part A Cohort 1d: Arm N3+RT | Part B Cohort 1c: Arm N3+RT+TMZ | Part B Cohort 1d: Arm N3+RT
Number analyzed (Participants) | 10 | 10 | 20 | 31 | 30 | 28 | 28
Percentage of participants
  Grade 1 | 0 | 0 | 0 | 3.2 | 0 | 0 | 0
  Grade 2 | 0 | 10.0 | 5.0 | 0 | 16.7 | 3.6 | 10.7
  Grade 3 | 60.0 | 40.0 | 35.0 | 45.2 | 16.7 | 35.7 | 32.1
  Grade 4 | 20.0 | 0 | 15.0 | 16.1 | 16.7 | 3.6 | 14.3
  Grade 5 | 0 | 0 | 0 | 0 | 3.3 | 3.6 | 0

4. Primary Outcome: Percentage of Participants With Specific Laboratory Abnormalities in Liver Tests in Cohorts 1, 1b, 1c and 1d
Description: The percentage of participants who experienced a laboratory abnormality of the liver in each treatment arm.
  MedDRA Version: 24.1
  Aspartate aminotransferase (AST) Alanine aminotransferase (ALT) Upper Limit of Normal (ULN) Denominator corresponds to participants with at least on one treatment measurement of the corresponding laboratory parameter. Includes laboratory results reported after the first dose and within 30 days of last dose of study therapy.
Time Frame: From first dose to 30 days post last dose (up to approximately 34 months).
Population: All Treated Subjects in Cohorts 1, 1b, 1c and 1d with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Arm N1+I3 | Cohort 1: Arm N3 | Cohort 1b: Arm N3+I1 | Part A Cohort 1c: Arm N3+RT+TMZ | Part A Cohort 1d: Arm N3+RT | Part B Cohort 1c: Arm N3+RT+TMZ | Part B Cohort 1d: Arm N3+RT
Number analyzed (Participants) | 10 | 10 | 19 | 31 | 30 | 27 | 27
Percentage of participants
  ALT OR AST > 3*ULN | 30.0 | 0.0 | 15.8 | 22.6 | 10.0 | 18.5 | 14.8
  ALT OR AST > 5*ULN | 20.0 | 0.0 | 10.5 | 12.9 | 3.3 | 11.1 | 3.7
  ALT OR AST > 10*ULN | 10.0 | 0.0 | 5.3 | 6.5 | 3.3 | 3.7 | 3.7
  ALT OR AST > 20*ULN | 10.0 | 0.0 | 5.3 | 3.2 | 3.3 | 0.0 | 3.7
  TOTAL BILIRUBIN (Tbili) > 2*ULN | 10.0 | 0.0 | 0.0 | 0.0 | 0.0 | 7.4 | 0.0
  ALP > 1.5*ULN | 10.0 | 10.0 | 0.0 | 0.0 | 3.3 | 0.0 | 3.7
  ALT or AST > 3xULN w/ Tbili > 1.5*ULN within 1 day | 10.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.7 | 0.0
  ALT or AST > 3*ULN w/ Tbili > 1.5*ULN within 30 days | 10.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.7 | 0.0
  ALT or AST > 3xULN w/ Tbili > 2*ULN within 1 day | 10.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.7 | 0.0
  ALT or AST > 3*ULN w/ Tbili > 2*ULN within 30 days | 10.0 | 0.0 | 0.0 | 0.0 | 0.0 | 3.7 | 0.0

5. Primary Outcome: Percentage of Participants With Specific Laboratory Abnormalities in Thyroid Tests in Cohorts 1, 1b, 1c and 1d
Description: The percentage of participants who experienced a laboratory abnormality of the thyroid in each treatment arm.
  MedDRA Version: 24.1
  Free T3 (FT3) Free T4 (FT4) Lower Limit of Normal (LLN)
  (A) Within a 2-week window after the abnormal TSH test date. (B) Includes participants with TSH abnormality and with no FT3/FT4 test values in the 2-week window or with non-abnormal value(s) from only one of the two tests and no value from the other test.
Time Frame: From first dose to 30 days post last dose (up to approximately 34 months).
Population: All Treated Subjects in Cohorts 1, 1b, 1c and 1d with at Least One On-Treatment TSH measurement
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Arm N1+I3 | Cohort 1: Arm N3 | Cohort 1b: Arm N3+I1 | Part A Cohort 1c: Arm N3+RT+TMZ | Part A Cohort 1d: Arm N3+RT | Part B Cohort 1c: Arm N3+RT+TMZ | Part B Cohort 1d: Arm N3+RT
Number analyzed (Participants) | 10 | 10 | 19 | 30 | 30 | 27 | 27
Percentage of participants
  TSH > ULN | 20.0 | 50.0 | 10.5 | 23.3 | 16.7 | 11.1 | 7.4
  TSH > ULN, WITH TSH <= ULN AT BASELINE | 20.0 | 30.0 | 10.5 | 20.0 | 16.7 | 11.1 | 7.4
  TSH > ULN, WITH AT LEAST ONE FT3/FT4 TEST < LLN | 20.0 | 30.0 | 10.5 | 13.3 | 13.3 | 7.4 | 0.0
  TSH > ULN, WITH ALL OTHER FT3/FT4 TEST >= LLN | 0.0 | 10.0 | 0.0 | 6.7 | 0.0 | 3.7 | 7.4
  TSH > ULN, WITH FT3/FT4 TEST MISSING | 0.0 | 10.0 | 0.0 | 3.3 | 3.3 | 0.0 | 0.0
  TSH < LLN | 60.0 | 30.0 | 31.6 | 43.3 | 40.0 | 22.2 | 33.3
  TSH < LLN, WITH TSH >= LLN AT BASELINE | 60.0 | 30.0 | 31.6 | 33.3 | 40.0 | 18.5 | 18.5
  TSH<LLN, LLN WITH AT LEAST ONE FT3/FT4 TEST>ULN | 30.0 | 10.0 | 15.8 | 10.0 | 13.3 | 11.1 | 0.0
  TSH < LLN, WITH ALL OTHER FT3/FT4 TEST <= ULN | 20.0 | 20.0 | 10.5 | 30.0 | 16.7 | 11.1 | 29.6
  TSH < LLN, WITH FT3/FT4 TEST MISSING | 10.0 | 0.0 | 5.3 | 3.3 | 10.0 | 0.0 | 3.7

6. Primary Outcome: Overall Survival (OS) for Cohort 2
Description: OS was measured in months from the time of randomization to the event date (death) due to any cause. A participant who has not died will be censored at the last known alive date.
  Based on Kaplan-Meier Estimates. Hazard ratio from Cox proportional hazard model stratified by presence of measurable lesions at baseline per IVRS. P-value from log-rank test stratified by presence of measurable lesions at baseline per IVRS.
Time Frame: Time between the date of randomization and the date of death due to any cause (up to up to 17Jun2019, approximately 5 years)
Population: All Randomized Participants in Cohort 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2: Arm N3 | Cohort 2: Arm B
Number analyzed (Participants) | 184 | 185
Months | 9.77 [8.21 to 11.83] | 10.05 [9.00 to 11.99]
Statistical Analysis 1: Comparison: Cohort 2: Arm N3 vs Cohort 2: Arm B; Test type: Superiority; p = 0.3791, log-rank test stratified; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.89 to 1.36]

7. Secondary Outcome: Overall Survival (OS) at 12 Months for Cohort 2
Description: OS(12) is measured as the percentage of participants alive at 12 months per Kaplan-Meier curve of OS. Z test with variance estimation based on Greenwood formula using log(-log) transformation.
Time Frame: From randomization to 12 months following randomization
Population: All Randomized Participants in Cohort 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 2: Arm N3 | Cohort 2: Arm B
Number analyzed (Participants) | 184 | 185
Percentage of Participants | 41.8 [34.7 to 48.8] | 42.4 [34.9 to 49.6]
Statistical Analysis 1: Comparison: Cohort 2: Arm N3 vs Cohort 2: Arm B; Test type: Superiority; p = 0.9208, Z test with variance estimation based on; Greenwood formula using log(-log) transformation; Difference of OS rates at 12 months = -0.5, 95% CI 2-sided [-10.8 to 9.7]

8. Secondary Outcome: Overall Survival (OS) for Cohorts 1c and 1d
Description: OS was measured in months from the time of randomization (Part B) or time of treatment (Part A) to the event date (death) due to any cause. A participant who has not died will be censored at the last known alive date.
  Based on Kaplan-Meier Estimates.
Time Frame: Time between the date of randomization and the date of death due to any cause (up to approximately 10 years and 5 months)
Population: All Randomized (Part B) or Treated (Part A) Participants in Cohorts 1c and 1d
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A Cohort 1c: Arm N3+RT+TMZ | Part A Cohort 1d: Arm N3+RT | Part B Cohort 1c: Arm N3+RT+TMZ | Part B Cohort 1d: Arm N3+RT
Number analyzed (Participants) | 31 | 30 | 28 | 28
Months | 22.08 [16.13 to 32.39] | 14.41 [12.55 to 17.31] | 15.95 [10.35 to 18.30] | 13.96 [10.81 to 18.14]

9. Secondary Outcome: Progression Free Survival (PFS) for Cohort 2
Description: PFS was measured in months from the time of randomization to the date of the first documented tumor progression or death due to any cause. Based on Kaplan-Meier Estimates. Hazard ratio from Cox proportional hazard model stratified by presence of measurable lesions at baseline per IVRS.
Time Frame: Time from randomization to the date of the first documented tumor progression or death due to any cause (up to approximately 10 years and 5 months)
Population: All Randomized Participants in Cohort 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2: Arm N3 | Cohort 2: Arm B
Number analyzed (Participants) | 184 | 185
Months | 1.51 [1.48 to 1.61] | 3.61 [2.99 to 4.60]
Statistical Analysis 1: Comparison: Cohort 2: Arm N3 vs Cohort 2: Arm B; Test type: Superiority; Hazard Ratio (HR) = 1.88, 95% CI 2-sided [1.50 to 2.35]

10. Secondary Outcome: Objective Response Rate (ORR) for Cohort 2
Description: ORR was measured by the percentage of participants whose best overall response (BOR) is confirmed Complete Response (CR) or Partial Response (PR) divided by response evaluable participants. The best overall response (BOR) is determined once all the data for the participant is known. BOR is defined as the best response designation, as determined by investigators, recorded between the date of randomization and the date of objectively documented progression per RANO criteria, the date of subsequent therapy, or date of surgical resection, whichever occurs first.
  Confidence interval based on the Clopper and Pearson method. For the comparison of the odds ratio of Nivolumab over Bevacizumab, the Cochran-Mantel-Haenszel (CMH) method of weighting was utilized.
Time Frame: as for outcome 9
Population: All Response Evaluable Participants in Cohort 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 2: Arm N3 | Cohort 2: Arm B
Number analyzed (Participants) | 153 | 156
Percentage of participants | 7.8 [4.1 to 13.3] | 23.1 [16.7 to 30.5]
Statistical Analysis 1: Comparison: Cohort 2: Arm N3 vs Cohort 2: Arm B; Test type: Superiority; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.15 to 0.59]

11. Post Hoc Outcome: Overall Survival (OS) for Cohort 2 - Extended Collection
Description: as for outcome 6
Time Frame: as for outcome 8
Population: All Randomized Participants in Cohort 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2: Arm N3 | Cohort 2: Arm B
Number analyzed (Participants) | 184 | 185
Months | 9.77 [8.21 to 11.83] | 10.05 [9.00 to 11.99]
Statistical Analysis 1: Comparison: Cohort 2: Arm N3 vs Cohort 2: Arm B; Test type: Superiority; p = 0.3791, log-rank test stratified; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.89 to 1.36]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From randomization (cohorts 1, 2, and 1c/1d of Part B) or first dose (cohorts 1b, and 1c/1d of Part A) through the course of the trial (up to approximately 125 months). SAEs and NSAEs: From first dose (SAEs and NSAEs) to 100 days post last dose (up to approximately 113 months). SAEs = Serious Adverse Events NSAEs = Non-Serious Adverse Events ("Other Adverse Events", as labeled in the table below)
Description: All-Cause Mortality = randomized (cohorts 1, 2, and 1c/1d of Part B) and treated (cohorts 1b, and 1c/1d of Part A) participant populations.
  SAEs and NSAEs (Other Adverse Events) = treated participant population
Arm/Group | Cohort 1: Arm N1+I3 | Cohort 1: Arm N3 | Cohort 1b: Arm N3+I1 | Part A Cohort 1c: Arm N3+RT+TMZ | Part A Cohort 1d: Arm N3+RT | Part B Cohort 1c: Arm N3+RT+TMZ | Part B Cohort 1d: Arm N3+RT | Cohort 2: Arm N3 | Cohort 2: Arm B
All-Cause Mortality (participants affected / at risk) | 10/10 | 9/10 | 20/20 | 29/31 | 30/30 | 28/29 | 28/30 | 180/184 | 166/185
Serious Adverse Events (participants affected / at risk) | 8/10 | 7/10 | 15/20 | 24/31 | 19/30 | 16/28 | 19/28 | 117/182 | 94/165
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 20/20 | 31/31 | 29/30 | 27/28 | 27/28 | 168/182 | 148/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Arm N1+I3 (N=10) | Cohort 1: Arm N3 (N=10) | Cohort 1b: Arm N3+I1 (N=20) | Part A Cohort 1c: Arm N3+RT+TMZ (N=31) | Part A Cohort 1d: Arm N3+RT (N=30) | Part B Cohort 1c: Arm N3+RT+TMZ (N=28) | Part B Cohort 1d: Arm N3+RT (N=28) | Cohort 2: Arm N3 (N=182) | Cohort 2: Arm B (N=165)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye movement disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Necrosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 4 | 1 | 1 | 2 | 3 | 2
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalitis herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Graft infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes simplex encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 5 | 0 | 1 | 3 | 4 | 2
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 3 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza B virus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 8 | 12 | 9 | 4 | 7 | 64 | 53
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 3 | 2 | 3 | 2 | 2 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 5 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Demyelination (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 2 | 0 | 5 | 1 | 10 | 2
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 5 | 3
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 1 | 5 | 4 | 4 | 2 | 17 | 11
Slow speech (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 2 | 2 | 4 | 3 | 1 | 1 | 3 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Granulomatous pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 4 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 5
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Arm N1+I3 (N=10) | Cohort 1: Arm N3 (N=10) | Cohort 1b: Arm N3+I1 (N=20) | Part A Cohort 1c: Arm N3+RT+TMZ (N=31) | Part A Cohort 1d: Arm N3+RT (N=30) | Part B Cohort 1c: Arm N3+RT+TMZ (N=28) | Part B Cohort 1d: Arm N3+RT (N=28) | Cohort 2: Arm N3 (N=182) | Cohort 2: Arm B (N=165)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 7 | 1 | 2 | 4 | 8 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 1 | 2 | 0 | 6 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 2 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 3
Cushingoid (Endocrine disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2
Endocrine disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 1 | 1 | 2 | 3 | 0 | 0 | 5 | 0
Hypothyroidism (Endocrine disorders) | 1 | 2 | 1 | 3 | 3 | 2 | 3 | 9 | 2
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 2 | 2 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0
Night blindness (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 6 | 3 | 1 | 0 | 5 | 4
Visual field defect (Eye disorders) | 0 | 1 | 1 | 3 | 0 | 2 | 0 | 3 | 3
Visual impairment (Eye disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 3 | 4 | 3 | 2 | 3 | 17 | 5
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 4 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 4 | 10 | 4 | 12 | 1 | 26 | 15
Diarrhoea (Gastrointestinal disorders) | 7 | 2 | 7 | 8 | 4 | 3 | 8 | 28 | 16
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 9 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 5 | 4
Nausea (Gastrointestinal disorders) | 3 | 3 | 6 | 13 | 8 | 15 | 7 | 27 | 22
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 6
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 4 | 4
Vomiting (Gastrointestinal disorders) | 4 | 2 | 4 | 6 | 3 | 7 | 3 | 15 | 11
Asthenia (General disorders) | 0 | 1 | 2 | 1 | 1 | 3 | 1 | 14 | 9
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Chills (General disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 3 | 2
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 8 | 5 | 14 | 25 | 16 | 20 | 18 | 69 | 45
Gait disturbance (General disorders) | 3 | 2 | 6 | 5 | 3 | 2 | 0 | 16 | 7
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 2 | 5
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 4
Oedema (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 2 | 0 | 2 | 4 | 2 | 0 | 2 | 16 | 15
Pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 5 | 2 | 4 | 5
Pyrexia (General disorders) | 2 | 0 | 2 | 3 | 3 | 3 | 6 | 13 | 8
Candida infection (Infections and infestations) | 2 | 0 | 2 | 1 | 3 | 2 | 3 | 1 | 4
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 7 | 6
Oral candidiasis (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 5 | 2
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 2
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 4 | 1 | 1 | 1 | 6 | 6
Urinary tract infection (Infections and infestations) | 0 | 0 | 5 | 1 | 2 | 1 | 2 | 11 | 7
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 4 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 5 | 3 | 3 | 2 | 1 | 18 | 10
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 3 | 9 | 5 | 5 | 2 | 16 | 10
Amylase increased (Investigations) | 3 | 1 | 1 | 4 | 2 | 2 | 2 | 4 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 2 | 9 | 3 | 4 | 2 | 6 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 5 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 3 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 3 | 2
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Lipase increased (Investigations) | 4 | 2 | 2 | 6 | 5 | 2 | 1 | 10 | 5
Lymphocyte count decreased (Investigations) | 0 | 0 | 3 | 6 | 3 | 3 | 2 | 2 | 5
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 5 | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 3 | 8 | 2 | 5 | 2 | 7 | 5
Weight decreased (Investigations) | 0 | 0 | 1 | 4 | 3 | 1 | 3 | 5 | 7
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 5 | 4
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 6 | 1 | 2 | 1 | 2 | 3
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 3 | 5 | 3 | 7 | 9 | 11 | 9
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2 | 3 | 1 | 0 | 4 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 5 | 7 | 7 | 6 | 2 | 10 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 2
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 4 | 2 | 2 | 2 | 5 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 5 | 5 | 2 | 2 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 9 | 4 | 7 | 4 | 26 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 6 | 2 | 1 | 5 | 13 | 11
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 10 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5 | 3 | 2 | 3 | 3 | 15 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3 | 1 | 3 | 0 | 7 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 6 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 15 | 9
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 4 | 3
Aphasia (Nervous system disorders) | 0 | 0 | 2 | 6 | 3 | 5 | 3 | 28 | 21
Ataxia (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 5 | 2
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 7 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 8 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1 | 3 | 5 | 2 | 1 | 3 | 10 | 6
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 9 | 2
Dizziness (Nervous system disorders) | 1 | 4 | 4 | 8 | 5 | 2 | 3 | 16 | 11
Dysarthria (Nervous system disorders) | 1 | 2 | 2 | 2 | 1 | 0 | 4 | 5 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 0
Dyspraxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 2
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 7 | 7 | 10 | 14 | 13 | 17 | 11 | 57 | 53
Hemiparesis (Nervous system disorders) | 3 | 3 | 7 | 5 | 2 | 4 | 3 | 27 | 16
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 5 | 1 | 1 | 5 | 5
Lethargy (Nervous system disorders) | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 3 | 4 | 2 | 3 | 1 | 1 | 14 | 10
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 3 | 1 | 3 | 2 | 9 | 5
Partial seizures (Nervous system disorders) | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 5 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Psychomotor skills impaired (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 2
Seizure (Nervous system disorders) | 1 | 2 | 2 | 3 | 7 | 6 | 12 | 33 | 17
Syncope (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1 | 2 | 3 | 1 | 2 | 4 | 4
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 5 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 2 | 4 | 5 | 1 | 4 | 6 | 6
Confusional state (Psychiatric disorders) | 3 | 3 | 9 | 2 | 3 | 6 | 3 | 15 | 10
Delusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 1 | 3 | 6 | 1 | 6 | 10
Disorientation (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 3
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 2 | 5 | 6 | 3 | 16 | 15
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 3
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 12
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 4 | 1 | 3 | 1 | 1 | 8 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 9 | 5 | 5 | 3 | 5 | 23 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3 | 1 | 1 | 2 | 5 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 4 | 2 | 2 | 3 | 7 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 0 | 3 | 0 | 7 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 2
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 5 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6 | 2 | 4 | 5 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 3 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 8 | 1 | 0 | 3 | 13 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 6 | 7 | 3 | 2 | 4 | 20 | 7
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 5 | 8 | 2 | 2 | 9 | 18 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 5 | 4 | 1 | 1 | 7 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1 | 5 | 6 | 3 | 1 | 12 | 50
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 3 | 2
Pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT02017717/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT02017717/SAP_001.pdf